CLINICAL TRIAL: NCT03851523
Title: AlfaCognition: Longitudinal Study for the Characterization of the Phases of Subjective Perception of Cognitive Decline and Mild Cognitive Impairment of Alzheimer's Disease.
Brief Title: Longitudinal Study for the Characterization of the Phases of Subjective Perception of Cognitive Decline and Mild Cognitive Impairment of Alzheimer's Disease.
Status: Recruiting | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ALFAcognition/BBRC2017
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Subjective Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood for subsequent DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Alzheimer's disease (AD) is the leading cause of dementia and its prevalence is estimated to exceed 100 million affects by 2050, becoming the main public health problem worldwide. AD is considered a clinicopathological entity characterized by a progressive cognitive impairment with affectation of memory and other cognitive domains, which underlies a neuropathological pattern with extracellular accumulation of β-amyloid protein (Aβ) in the form of neuritic plaques, intracellular deposits of tau protein in the form of neuritic strands and neurofibrillary tangles, neuronal and synaptic loss and glial proliferation. Classically, its definitive diagnosis implied the existence of a clinical phenotype compatible with dementia, together with the neuropathological findings characteristic of the disease. More recently, evidence of clinical and biological changes leading to the dementia phase has led to the development of new diagnostic criteria that divide the course of AD into 3 stages: (1) a pre-clinical phase, which would include persons with positive biomarkers with normal cognitive performance for their age and educational level; (2) a phase of mild cognitive impairment (MCI), characterized by cognitive performance lower than expected by age and educational level; and (3) a dementia phase, once cognitive deficits interfere with the activities of daily living.

Recent research has also shed light into the subdivision of each of the above-mentioned stages in distinct phases. For example, the existence of a subjective perception of cognitive decline or a subtle cognitive decline, have been postulated as phases within the AD preclinical stage.

The lack of positive results in the different clinical trials performed to date in patients with AD dementia has redirected the focus of therapeutic strategies towards preventing the development of dementia. For this reason, a detailed characterization of the successive clinical and biological changes that lead to the dementia stage is of vital importance in identifying the persons who could benefit from a possible preventive strategy, as well as the optimal moment to carry out the intervention. The the scientific community, is convinced that intervention aiming to prevent the clinical development of AD dementia must be implemented several years before the first symptoms arise.

In this context, the present project is developed under the hypothesis that subjective cognitive decline (SCD) in individuals with a performance in cognitive tests within normality represents the first symptomatic manifestation of AD. In persons with SCD, the presence of a higher intensity of subjective complaint quantified using a specific subjective complaint questionnaire (SCD-Q) will be associated with lower cognitive performance and a higher rate of conversion to MCI and/or dementia. The relationship between the perception of cognitive decline by the subject and his/her relative will differently vary depending on the stage of the disease: in subjects with progressive cognitive impairment, the subjective perception of cognitive decline will decrease with disease progression whereas the perception of decline will increase with disease progression in their relatives. The degree of perception of cognitive decline throughout the different phases of the disease will be correlated with cognitive and affective patterns as well as with changes in AD biomarkers. These changes will be related to specific brain patterns and abnormal levels of AD biomarkers, which on the other hand will also be present in patients with MCI and mild dementia due to AD.

The present study has two main objectives that are:

1. To characterize from a cognitive and biomarker (when available) point of view persons with SCD and to study its association with the risk of presenting a progressive cognitive deterioration.
2. To study the evolution of the subjective perception of cognitive impairment by the participants and their relatives and to analyze its impact in cognitive, affective and functional terms along the clinical-biological continuum of AD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 45 and 74 years at the time of inclusion in the 45-65/FPM2012 study or older than 45 for persons who have not previously participated in 45-65/FPM2012.
2. Cognitively healthy persons with SCD, as well as people with MCI and mild dementia.
3. Participation of a relative to perform the subjective memory complaint and clinical interview.

Exclusion criteria:

1. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol.
2. Any significant disorder that could course with cognitive impairment that is not related to AD.
3. Family history of monogenic AD.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cognitively unimpaired subjects with SCD or MCI/mild dementia individuals
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive Decline Questionnaire (my-Cog) | at inclusion
  Change in my-Cog score between groups - total score 0-24
Subjective Cognitive Decline Questionnaire (their-Cog) | at inclusion
  Change in their-Cog score between groups - total score 0-24

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No